CLINICAL TRIAL: NCT04381676
Title: The Flipped Classroom Approach to Teaching Horizontal Strabismus in Ophthalmology Residency: A Multi-Centered Randomized Controlled Study
Brief Title: The Flipped Classroom Approach in Ophthalmology Residency
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Michelle T. Cabrera, Associate Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00001185
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Educational Problems
Keywords: Flipped Classroom

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flipped Classroom: Residents in the flipped classroom were assigned a pre-class video lecture prior to completing the flipped classroom in-class case-based activity in groups of 2-3 each.
  Interventions: Other: Flipped Classroom Approach
- Traditional Classroom: Residents in the traditional classroom were assigned a pre-class reading assignment followed by a 44-minute lecture that was delivered in-person using PowerPoint.

INTERVENTIONS:
Other: Flipped Classroom Approach — In the Flipped Classroom, participants form groups of 2-3 and are instructed to work together through clinical cases of the in-class case based activity, committing to group answers to the clinical questions before advancing to the next case. At the end of class, the faculty instructor facilitated a short interactive group discussion.
  Groups: Flipped Classroom

SUMMARY:
This study aims to evaluate the flipped classroom approach compared to the traditional classroom approach in teaching horizontal strabismus in ophthalmology residency didactics.

DETAILED DESCRIPTION:
Ophthalmology residents (post-graduate years 2-4) from 11 institutions were invited to participate. Participating residents were taught esotropia and exotropia topics sequentially, randomized by order and classroom style (flipped classroom vs. traditional lecture) one to three weeks apart. Participants were assigned a pre-class video lecture prior to the flipped classroom in-class case-based activity. The traditional classroom included a preparatory reading assignment and an in-person lecture delivered by the same instructor. Participants completed three identical 5-question content assessments (pre-test, post-test, and 3-month retention) and opinion surveys following each classroom.

ELIGIBILITY:
Inclusion Criteria:

* Ophthalmology residents of all levels (PGY2-PGY4) from 11 residency programs were invited to participate in this study

Exclusion Criteria:

* Those who did not complete both classroom styles were excluded from the survey data
* Those who lost their study-IDs were excluded from the results analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ophthalmology residents from all levels (PGY2-PGY4) in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Resident Preference | Through study completion, an average of 2 weeks
  Participants were asked to complete both a written (Likert-scale) survey in the classroom and an additional online survey (Catalyst WebQ, University of Washington, Seattle, WA) following the classroom session. These surveys asked residents to rate their preference for traditional vs. flipped classroom format, the effectiveness of preparation and classroom material, and the advantages and disadvantages of the flipped classroom format

SECONDARY OUTCOMES:
Knowledge Acquisition | Baseline (Before class), immediately after completing the class, 3 months after class
  Participants were assessed a total of three times for each course (esotropia and exotropia): once prior to starting the class (pre-test), once immediately after completing the class (post-test), and once three months later. All assessments consisted of 5 OKAP style questions created by fellowship trained ophthalmologists. These test questions were previously piloted. Residents were allotted 5 minutes to complete each test.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle T Cabrera, MD, Principal Investigator — University of Washington
Locations (1):
- Department of Ophthalmology - University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krathwohl, D. R. (2002). A revision of Bloom's taxonomy: an overview. Theory into practice, 41(4), 212-218.
- [Background] Cabrera MT, Yanovitch TL, Gandhi NG, Ding L, Enyedi LB. The flipped-classroom approach to teaching horizontal strabismus in ophthalmology residency: a pilot study. J AAPOS. 2019 Aug;23(4):200.e1-200.e6. doi: 10.1016/j.jaapos.2019.02.009. Epub 2019 Jun 20. PMID 31229609
- [Background] Casasola T SK, Nguyen T, Warschauer M. Can flipping the classroom work? Evidence from undergraduate chemistry. International Journal of Teaching and Learning in Higher Education. 2017;29(3):421-435.
- [Background] Baepler PM WJ, Driessen M. It's not about seat time: Blending, flipping, and efficiency in active learning classrooms. Computers & Education. 2014;78:227-236.
- [Background] O'Flaherty J PC. The use of flipped classrooms in higher education: A scoping review. The Internet and Higher Education. 2015;25:85-95.
- [Background] Nouri, J. The flipped classroom: for active, effective and increased learning - especially for low achievers. Int J Educ Technol High Educ 13, 33 (2016).
- [Background] Soriano RP, Blatt B, Coplit L, CichoskiKelly E, Kosowicz L, Newman L, Pasquale SJ, Pretorius R, Rosen JM, Saks NS, Greenberg L. Teaching medical students how to teach: a national survey of students-as-teachers programs in U.S. medical schools. Acad Med. 2010 Nov;85(11):1725-31. doi: 10.1097/ACM.0b013e3181f53273. PMID 20881824
- [Background] Yu TC, Wilson NC, Singh PP, Lemanu DP, Hawken SJ, Hill AG. Medical students-as-teachers: a systematic review of peer-assisted teaching during medical school. Adv Med Educ Pract. 2011 Jun 23;2:157-72. doi: 10.2147/AMEP.S14383. Print 2011. PMID 23745087
- [Background] Freeman S, Eddy SL, McDonough M, Smith MK, Okoroafor N, Jordt H, Wenderoth MP. Active learning increases student performance in science, engineering, and mathematics. Proc Natl Acad Sci U S A. 2014 Jun 10;111(23):8410-5. doi: 10.1073/pnas.1319030111. Epub 2014 May 12. PMID 24821756
- [Background] Wolff M, Wagner MJ, Poznanski S, Schiller J, Santen S. Not another boring lecture: engaging learners with active learning techniques. J Emerg Med. 2015 Jan;48(1):85-93. doi: 10.1016/j.jemermed.2014.09.010. Epub 2014 Oct 13. PMID 25440868
- [Background] Young TP, Bailey CJ, Guptill M, Thorp AW, Thomas TL. The flipped classroom: a modality for mixed asynchronous and synchronous learning in a residency program. West J Emerg Med. 2014 Nov;15(7):938-44. doi: 10.5811/westjem.2014.10.23515. Epub 2014 Oct 29. PMID 25493157
- [Background] Riddell J, Jhun P, Fung CC, Comes J, Sawtelle S, Tabatabai R, Joseph D, Shoenberger J, Chen E, Fee C, Swadron SP. Does the Flipped Classroom Improve Learning in Graduate Medical Education? J Grad Med Educ. 2017 Aug;9(4):491-496. doi: 10.4300/JGME-D-16-00817.1. PMID 28824764
- [Background] Martinelli SM, Chen F, DiLorenzo AN, Mayer DC, Fairbanks S, Moran K, Ku C, Mitchell JD, Bowe EA, Royal KD, Hendrickse A, VanDyke K, Trawicki MC, Rankin D, Guldan GJ, Hand W, Gallagher C, Jacob Z, Zvara DA, McEvoy MD, Schell RM. Results of a Flipped Classroom Teaching Approach in Anesthesiology Residents. J Grad Med Educ. 2017 Aug;9(4):485-490. doi: 10.4300/JGME-D-17-00128.1. PMID 28824763
- [Background] Marchalot A, Dureuil B, Veber B, Fellahi JL, Hanouz JL, Dupont H, Lorne E, Gerard JL, Compere V. Effectiveness of a blended learning course and flipped classroom in first year anaesthesia training. Anaesth Crit Care Pain Med. 2018 Oct;37(5):411-415. doi: 10.1016/j.accpm.2017.10.008. Epub 2017 Nov 22. PMID 29175318
- [Background] Allenbaugh J, Spagnoletti C, Berlacher K. Effects of a Flipped Classroom Curriculum on Inpatient Cardiology Resident Education. J Grad Med Educ. 2019 Apr;11(2):196-201. doi: 10.4300/JGME-D-18-00543.1. PMID 31024653
- [Background] Bachorik A, Nemer MK, Chen GL, Alexander CB, Pelletier SR, Pace LE, Shields HM. Case-Based Curriculum With Integrated Smartphone Applications Improves Internal Medicine Resident Knowledge Of Contraceptive Care. Adv Med Educ Pract. 2019 Nov 19;10:971-977. doi: 10.2147/AMEP.S221256. eCollection 2019. PMID 31819696
- [Background] Moulton ST, Turkay S, Kosslyn SM. Does a presentation's medium affect its message? PowerPoint, Prezi, and oral presentations. PLoS One. 2017 Jul 5;12(7):e0178774. doi: 10.1371/journal.pone.0178774. eCollection 2017. PMID 28678855
- [Background] Låg, T., & Sæle, R. G. (2019). Does the Flipped Classroom Improve Student Learning and Satisfaction? A Systematic Review and Meta-Analysis. AERA Open.
- [Background] Hew KF, Lo CK. Flipped classroom improves student learning in health professions education: a meta-analysis. BMC Med Educ. 2018 Mar 15;18(1):38. doi: 10.1186/s12909-018-1144-z. PMID 29544495